CLINICAL TRIAL: NCT02273050
Title: A Multicenter, Randomized, Double-Blind, Active-Controlled, Phase 3 Trial to Evaluate the Efficacy and Safety of Saxagliptin in Combination With Metformin IR as Initial Therapy Compared to Saxagliptin Monotherapy and to Metformin IR Monotherapy in Subjects With Type 2 Diabetes Who Have Inadequate Glycaemic Control
Brief Title: Evaluate the Efficacy and Safety of Saxagliptin in Combination With Metformin IR Compared to Saxagliptin Monotherapy and to Metformin IR Monotherapy in Drug Naive Chinese Subjects With Type 2 Diabetes Who Have Inadequate Glycaemic Control
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1680C00009
Record Dates: First submitted 2014-10-22; First posted 2014-10-23 (Estimated); Results first posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2017-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus, Dipeptidyl-Peptidase 4 Inhibitors, Saxagliptin, Metformin, Endocrine System Diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Endocrine System Diseases | interventions — saxagliptin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Saxagliptin 5 mg + Metformin (500 mg with titration) (Experimental): Saxagliptin 5 mg once daily and metformin 500 mg once daily, then titrate. Acarbose will be used as rescue medication as needed.
  Interventions: Drug: Saxagliptin 5 mg; Drug: Metformin 500 mg with titration
- Saxagliptin 5 mg + Placebo (Active Comparator): Saxagliptin 5 mg once daily and Placebo 500 mg once daily, then titrate. Acarbose will be used as rescue medication as needed.
  Interventions: Drug: Saxagliptin 5 mg; Drug: Placebo 500 mg for metformin (with titration)
- Metformin (500 mg with titration) + Placebo (Active Comparator): Placebo 5 mg once daily and metformin 500 mg once daily, then titrate. Acarbose will be used as rescue medication as needed.
  Interventions: Drug: Placebo 5 mg for Saxagliptin; Drug: Metformin 500 mg with titration

INTERVENTIONS:
Drug: Saxagliptin 5 mg — Tablet, Oral, 5 mg, Once daily in the morning
  Other Names: Onglyza; BMS-477118
  Arms: Saxagliptin 5 mg + Metformin (500 mg with titration); Saxagliptin 5 mg + Placebo
Drug: Placebo 5 mg for Saxagliptin — Tablet, Oral, 5 mg, Once daily in the morning
  Arms: Metformin (500 mg with titration) + Placebo
Drug: Placebo 500 mg for metformin (with titration) — Tablet, 500 mg, Once daily in the evening the first two weeks and thereafter according to titration.
  Arms: Saxagliptin 5 mg + Placebo
Drug: Metformin 500 mg with titration — Tablet, 500 mg, Once daily in the evening the first two weeks and thereafter according to titration.
  Other Names: Glucophage
  Arms: Metformin (500 mg with titration) + Placebo; Saxagliptin 5 mg + Metformin (500 mg with titration)

SUMMARY:
A Multicenter, Randomized, Double-Blind, Active-Controlled, Phase 3 Trial to Evaluate the Efficacy and Safety of Saxagliptin in Combination with Metformin IR as Initial Therapy Compared to Saxagliptin Monotherapy and to Metformin IR Monotherapy in Subjects with Type 2 Diabetes who have Inadequate Glycaemic Control

DETAILED DESCRIPTION:
Allocation: Randomized Endpoint Classification: Efficacy/Safety study Intervention Model: Parallel Assignment Masking: Double Blind Primary Purpose: Treatment

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with type 2 diabetes mellitus; 2. HbA1c ≥8% but ≤12%; 3.Fasting C-peptide ≥1.0 ng/ml; 4. Subject will be drug naïve; 5. Body mass index ≤40 kg/m2.

Exclusion Criteria:

1. Symptoms of poorly controlled diabetes; 2. Chronic or repeated intermittent corticosteroid treatment ; 3. Calculated creatinine clearance <60 ml/min or serum creatinine >132.6 μmol/L (>1.5 mg/dL) for men, >123.8 μmol/L (>1.4 mg/dL) for women; 4. Creatine Kinase ≥3x ULN; 5.Abnormal TSH value at screening will be further evaluated by free T4, subjects with an abnormal free T4 will be excluded; 6. History of administration of any antihyperglycaemic therapy for a total of 28 days or for more than three consecutive days or a total of seven non-consecutive days during the eight weeks prior to screening; 7. Current treatment with a strong CYP3A4/5 inhibitor; 8. Prior treatment with saxagliptin or any DPP-4 inhibitor; 9. Significant or history of cardiovascular disease, renal disease, psychiatric disorders, Immunocompromised individuals, hemoglobinopathies, liver disease, Pancreatitis.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1136 (Actual)
Dates: Start 2014-12; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Changyu Pan, Professor, Principal Investigator — The General Hospital of People's liberation Army
Locations (17):
- China (17):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Chuangchun
  - Research Site, Fuzhou
  - Research Site, Guiyang
  - Research Site, Hangzhou
  - Research Site, Ha’erbin
  - Research Site, Hefei
  - Research Site, Jinan
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Shijiazhuang
  - Research Site, Siping
  - Research Site, Tianjin
  - Research Site, Wuxi
  - Research Site, Yueyang

REFERENCES:
- [Derived] Dou J, Ma J, Liu J, Wang C, Johnsson E, Yao H, Zhao J, Pan C. Efficacy and safety of saxagliptin in combination with metformin as initial therapy in Chinese patients with type 2 diabetes: Results from the START study, a multicentre, randomized, double-blind, active-controlled, phase 3 trial. Diabetes Obes Metab. 2018 Mar;20(3):590-598. doi: 10.1111/dom.13117. Epub 2017 Oct 26. PMID 28926170

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 25 centers between 18 December 2014 and 03 August 2016.
Pre-assignment Details: The study duration was up to 27 weeks, consisting of an initial screening period lasting up to 2 weeks, a 1-week lead-in period, and a 24-week treatment period. The number of subjects who signed the ICF is 1136, the number of subjects randomized is 640.
Period: Overall Study
Arm/Group | METFORMIN + PLACEBO 5MG QD | SAXAGLIPTIN 5MG QD + METFORMIN | SAXAGLIPTIN 5MG QD + PLACEBO
Started | 210 | 216 | 214
Completed | 186 | 194 | 185
Not Completed | 24 | 22 | 29
Not completed — Adverse Event | 4 | 3 | 3
Not completed — Death | 0 | 0 | 1
Not completed — Dev. of study spec. withdrawal criteria | 0 | 1 | 1
Not completed — Lack of Efficacy | 0 | 1 | 1
Not completed — Withdrawal by Subject | 17 | 14 | 16
Not completed — Lost to Follow-up | 0 | 2 | 3
Not completed — Protocol Violation | 3 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | METFORMIN + PLACEBO 5MG QD | SAXAGLIPTIN 5MG QD + METFORMIN | SAXAGLIPTIN 5MG QD + PLACEBO | Total
Number analyzed (Participants) | 210 | 216 | 214 | 640
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.1 (11.08) [20 to 75] | 50.4 (10.78) [23 to 74] | 49.5 (10.93) [24 to 74] | 50.0 (10.92) [20 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 76 | 62 | 214
  Male | 134 | 140 | 152 | 426
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 210 | 216 | 214 | 640

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c From Baseline to Week 24 Provided That it is Prior to Rescue
Description: To evaluate the efficacy of the combination therapy (saxagliptin + metformin) when compared to placebo + metformin and placebo + saxagliptin with respect to reduction in HbA1c (%) at the end of 24 weeks of double-blinded treatment.
Time Frame: Baseline to Week 24 (prior to rescue)
Population: The full analysis set consisted of patients who were randomized, took at least 1 randomized study medication, and had both a baseline and at least 1 post-baseline efficacy assessment for the time point under consideration.
Measure: Least Squares Mean (Standard Error); unit: % HbA1c
Groups:
- Saxagliptin + Metformin: Saxagliptin 5 mg + Metformin 500 mg
- Saxagliptin + Placebo: Saxagliptin 5 mg + Placebo
- Metformin + Placebo: Metformin 500 mg + Placebo
Arm/Group | Saxagliptin + Metformin | Saxagliptin + Placebo | Metformin + Placebo
Number analyzed (Participants) | 209 | 212 | 204
% HbA1c | -3.007 (0.0706) [-3.146 to -2.869] | -2.123 (0.0701) [-2.260 to -1.985] | -2.794 (0.0715) [-2.935 to -2.654]
Statistical Analysis 1: Comparison: Saxagliptin + Metformin vs Saxagliptin + Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -0.885, 95% CI 2-sided [-1.080 to -0.689], Standard Error of Mean 0.0994
Statistical Analysis 2: Comparison: Saxagliptin + Metformin vs Metformin + Placebo; Test type: Superiority or Other; p = 0.034, ANCOVA; Mean Difference (Net) = -0.213, 95% CI 2-sided [-0.410 to -0.016], Standard Error of Mean 0.1005

2. Secondary Outcome: Glycemic Response Defined as HbA1c < 7.0% at Week 24
Description: To evaluate the efficacy of the combination therapy (saxagliptin + metformin) when compared to placebo + metformin and placebo + saxagliptin with respect to the proportion of subjects achieving a therapeutic glycemic response defined as HbA1c < 7.0% at the end of 24 weeks of double-blinded treatment.
Time Frame: Week 24 (prior to rescue)
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Saxagliptin + Metformin | Saxagliptin + Placebo | Metformin + Placebo
Number analyzed (Participants) | 209 | 212 | 204
Percentage of patients | 81.8 | 44.3 | 71.1
Statistical Analysis 1: Comparison: Saxagliptin + Metformin vs Saxagliptin + Placebo; Test type: Superiority or Other; p < 0.001, Fisher Exact; Mean Difference (Net) = 37.5, 95% CI 2-sided [29.0 to 46.0]
Statistical Analysis 2: Comparison: Saxagliptin + Metformin vs Metformin + Placebo; Test type: Superiority or Other; p = 0.011, Fisher Exact; Mean Difference (Net) = 10.7, 95% CI 2-sided [2.6 to 18.9]

3. Secondary Outcome: Change From Baseline to Week 24 (Prior to Rescue) in Fasting Plasma Glucose
Description: To evaluate the efficacy of the combination therapy (saxagliptin + metformin) when compared to placebo + metformin and placebo + saxagliptin with respect to reduction in fasting plasma glucose at the end of 24 weeks of double-blinded treatment.
Time Frame: Baseline to Week 24 prior to rescue
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Saxagliptin + Metformin | Saxagliptin + Placebo | Metformin + Placebo
Number analyzed (Participants) | 210 | 213 | 207
mmol/L | -3.25 (0.112) | -1.86 (0.111) | -2.94 (0.113)
Statistical Analysis 1: Comparison: Saxagliptin + Metformin vs Saxagliptin + Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -1.39, 95% CI 2-sided [-1.70 to -1.08], Standard Error of Mean 0.158
Statistical Analysis 2: Comparison: Saxagliptin + Metformin vs Metformin + Placebo; Test type: Superiority or Other; p = 0.046, ANCOVA; Mean Difference (Net) = -0.32, 95% CI 2-sided [-0.63 to 0.00], Standard Error of Mean 0.159

4. Secondary Outcome: Change From Baseline to Week 24 (Prior to Rescue) in Area Under the Curve From 0-180 Minutes for Postprandial Glucose Response to a Meal Tolerance Test
Description: To evaluate the efficacy of the combination therapy (saxagliptin + metformin) when compared to placebo + metformin and placebo + saxagliptin with respect to change in 180-minute postprandial glucose response to a meal tolerance test at the end of 24 weeks of double-blinded treatment.
Time Frame: Baseline to Week 24 prior to rescue
Population: The full analysis set consisted of patients who were randomized, took at least 1 randomized study medication, had both a baseline and at least 1 post-baseline efficacy assessment for the time point under consideration, and participated in a meal tolerance test.
Measure: Least Squares Mean (Standard Error); unit: mmol*min/L
Arm/Group | Saxagliptin + Metformin | Saxagliptin + Placebo | Metformin + Placebo
Number analyzed (Participants) | 120 | 117 | 113
mmol*min/L | -1027.8 (36.22) | -611.9 (36.69) | -858.5 (37.36)
Statistical Analysis 1: Comparison: Saxagliptin + Metformin vs Saxagliptin + Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -416.0, 95% CI 2-sided [-517.3 to -314.6], Standard Error of Mean 51.54
Statistical Analysis 2: Comparison: Saxagliptin + Metformin vs Metformin + Placebo; Test type: Superiority or Other; p = 0.001, ANCOVA; Mean Difference (Net) = -169.3, 95% CI 2-sided [-271.7 to -66.9], Standard Error of Mean 52.05

5. Secondary Outcome: Glycemic Response Defined as HbA1c ≤ 6.5% at Week 24
Description: To evaluate the efficacy of the combination therapy (saxagliptin + metformin) when compared to placebo + metformin and placebo + saxagliptin with respect to the proportion of subjects achieving a therapeutic glycemic response defined as HbA1c ≤ 6.5% at the end of 24 weeks of double-blinded treatment.
Time Frame: Week 24 (prior to rescue)
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Saxagliptin + Metformin | Saxagliptin + Placebo | Metformin + Placebo
Number analyzed (Participants) | 209 | 212 | 204
Percentage of patients | 67.0 | 32.1 | 55.4
Statistical Analysis 1: Comparison: Saxagliptin + Metformin vs Saxagliptin + Placebo; Test type: Superiority or Other; p < 0.001, Fisher Exact; Mean Difference (Net) = 34.9, 95% CI 2-sided [26.0 to 43.9]
Statistical Analysis 2: Comparison: Saxagliptin + Metformin vs Metformin + Placebo; Test type: Superiority or Other; p = 0.020, Fisher Exact; Mean Difference (Net) = 11.6, 95% CI 2-sided [2.3 to 20.9]

6. Secondary Outcome: Change From Baseline to Week 24 in 120-minute Postprandial Glucose Response to a Meal Tolerance Test
Description: To evaluate the efficacy of the combination therapy (saxagliptin + metformin) when compared to placebo + metformin and placebo + saxagliptin with respect to change in 120-minute postprandial glucose response to a meal tolerance test at the end of 24 weeks of double-blinded treatment.
Time Frame: Baseline to Week 24 prior to rescue
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Saxagliptin + Metformin | Saxagliptin + Placebo | Metformin + Placebo
Number analyzed (Participants) | 122 | 121 | 116
mmol/L | -7.09 (0.261) | -4.12 (0.262) | -5.95 (0.268)
Statistical Analysis 1: Comparison: Saxagliptin + Metformin vs Saxagliptin + Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -2.97, 95% CI 2-sided [-3.70 to -2.25], Standard Error of Mean 0.370
Statistical Analysis 2: Comparison: Saxagliptin + Metformin vs Metformin + Placebo; Test type: Superiority or Other; p = 0.002, ANCOVA; Mean Difference (Net) = -1.14, 95% CI 2-sided [-1.88 to -0.41], Standard Error of Mean 0.374

7. Secondary Outcome: Patients Rescued for Failing to Achieve Pre-specified Glycemic Targets or Discontinuation for Lack of Efficacy During the 24-week Double-blind Treatment Phase
Description: To evaluate the efficacy of the combination therapy (saxagliptin + metformin) when compared to placebo + metformin and placebo + saxagliptin with respect to the proportion of subjects requiring rescue for failing to achieve pre-specified glycemic targets or discontinuing for lack of efficacy within the 24 weeks of double-blinded treatment.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Saxagliptin + Metformin | Saxagliptin + Placebo | Metformin + Placebo
Number analyzed (Participants) | 210 | 213 | 207
Percentage of patients | 1.4 | 10.3 | 1.4
Statistical Analysis 1: Comparison: Saxagliptin + Metformin vs Saxagliptin + Placebo; Test type: Superiority or Other; p < 0.001, Fisher Exact; Mean Difference (Net) = -8.9, 95% CI 2-sided [-13.3 to -4.5]
Statistical Analysis 2: Comparison: Saxagliptin + Metformin vs Metformin + Placebo; Test type: Superiority or Other; p > 0.999, Fisher Exact; Mean Difference (Net) = 0.0, 95% CI 2-sided [-2.3 to 2.3]

ADVERSE EVENTS:
Description: Total number at risk is number of patients in safety analysis set (out of 640 randomized, 1 did not take study drug).
Arm/Group | METFORMIN + PLACEBO 5MG QD | SAXAGLIPTIN 5MG QD + METFORMIN | SAXAGLIPTIN 5MG QD + PLACEBO
Serious Adverse Events (participants affected / at risk) | 11/210 | 4/215 | 12/214
Other Adverse Events (participants affected / at risk) | 30/210 | 37/215 | 21/214
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | METFORMIN + PLACEBO 5MG QD (N=210) | SAXAGLIPTIN 5MG QD + METFORMIN (N=215) | SAXAGLIPTIN 5MG QD + PLACEBO (N=214)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatic mass (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatitis alcoholic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic hepatitis B (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Glomerulonephritis chronic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | METFORMIN + PLACEBO 5MG QD (N=210) | SAXAGLIPTIN 5MG QD + METFORMIN (N=215) | SAXAGLIPTIN 5MG QD + PLACEBO (N=214)
Diarrhoea (Gastrointestinal disorders) | 13 (19) | 14 (17) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 14 (14) | 15 (15) | 10 (11)
Hyperlipidaemia (Metabolism and nutrition disorders) | 7 (7) | 11 (11) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No